CLINICAL TRIAL: NCT02107261
Title: A Placebo-Controlled, Double-Blind, Randomized, Cross Over Pilot Study Of The Efficacy And Tolerability Of Incobotulinum Toxin A (Xeomin®) As A Treatment For Focal Task-Specific Dystonia Of The Musician's Hand
Brief Title: Incobotulinum Toxin A (Xeomin®) As A Treatment For Focal Task-Specific Dystonia Of The Musician's Hand
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Principal Investigator, David M. Simpson, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 13-1679
Record Dates: First submitted 2014-03-26; First posted 2014-04-08 (Estimated); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-04

CONDITIONS: Dystonia
Keywords: Musician's Dystonia
MeSH Terms: conditions — Dystonia; Dystonia, Focal, Task-Specific | interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Then Botulinum Toxin (Active Comparator): Placebo dose first does then boosters at week 2 and week 4 then 4 weeks washout, then Incobotulinumtoxin A first dose, with boosters at 2 week and week 4.
  Interventions: Drug: incobotulinumtoxin A; Drug: Placebo
- Incobotulinumtoxin A Then Placebo (Active Comparator): Incobotulinumtoxin A dose first does then boosters at week 2 and week 4 then 4 weeks washout, then Placebo first dose, with boosters at 2 week and week 4.
  Interventions: Drug: incobotulinumtoxin A; Drug: Placebo

INTERVENTIONS:
Drug: incobotulinumtoxin A — Incobotulinumtoxin A is being used on average doses between 10U and 30 Units per subject, but at no time will any subject receive over 100 Units. Each study visit, the assessing physician will select the muscles and the amounts of medication to be injected.
  Other Names: Xeomin
Drug: Placebo — matching placebo

SUMMARY:
The investigational drug being studied in this protocol is Incobotulinumtoxin A (Xeomin®). Botulinum toxin (BoNT) prevents the release of the acetylcholine from peripheral nerves, inhibiting muscle contractions. BoNT is effective in relaxing overactive muscles. In musician's dystonia, the ability to reduce abnormally overactive muscles in the hand can be critical for the musical professional to continue his or her career. With the use of EMG/electrical stimulation and/or ultrasound guidance, the injector can precisely localize the individual muscles that are affected in this condition with great accuracy. Prior studies have shown that BoNT injections produce beneficial effects in forearm muscles, and less effect in shoulder or proximal arm muscles.

Possible risks in treating patients with BoNT include excessive weakness of the injected muscles. The drug may also affect non-targeted muscles. However these risks will be minimized during the screening period by carefully targeting the affected muscles and by administering low doses of BoNT. Small booster doses may be given at follow up visit (2, 4, 14 and 16-weeks after the primary injection date) if the initial injection was insufficient to produce sufficient efficacy in relief of the focal dystonia and did not produce excess weakness of the targeted muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with focal task-specific dystonia of one or both hands, selectively triggered by performance on a musical instrument.
* Patients must have been evaluated by Dr. Frucht at the Movement Disorders Division of Mount Sinai Medical Center as part of their clinical care.
* Patients whose performance on an instrument is directly linked to their occupation.
* Patients must be between the ages of 18 and 80.
* Impairment in musical performance must be visible and demonstrable.

Exclusion Criteria:

* Patients whose dystonia is not severe enough to interfere with musical performance in the opinion of a skilled examiner.
* Patients with unstable medical conditions or psychiatric conditions.
* Patients with a medical condition that precludes them from receiving BoNT injections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Frucht, MD, Principal Investigator — NYU Langone Health; David M Simpson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Background] Jankovic J, Ashoori A. Movement disorders in musicians. Mov Disord. 2008 Oct 30;23(14):1957-65. doi: 10.1002/mds.22255. PMID 18785647
- [Background] Pullman SL, Hristova AH. Musician's dystonia. Neurology. 2005 Jan 25;64(2):186-7. doi: 10.1212/01.WNL.0000157497.08500.c1. No abstract available. PMID 15668411
- [Background] Altenmuller E. Focal dystonia: advances in brain imaging and understanding of fine motor control in musicians. Hand Clin. 2003 Aug;19(3):523-38, xi. doi: 10.1016/s0749-0712(03)00043-x. PMID 12945651
- [Background] Frucht SJ, Fahn S, Greene PE, O'Brien C, Gelb M, Truong DD, Welsh J, Factor S, Ford B. The natural history of embouchure dystonia. Mov Disord. 2001 Sep;16(5):899-906. doi: 10.1002/mds.1167. PMID 11746620
- [Background] Elbert T, Pantev C, Wienbruch C, Rockstroh B, Taub E. Increased cortical representation of the fingers of the left hand in string players. Science. 1995 Oct 13;270(5234):305-7. doi: 10.1126/science.270.5234.305. PMID 7569982
- [Background] Munte TF, Altenmuller E, Jancke L. The musician's brain as a model of neuroplasticity. Nat Rev Neurosci. 2002 Jun;3(6):473-8. doi: 10.1038/nrn843. PMID 12042882
- [Background] Altenmuller E, Baur V, Hofmann A, Lim VK, Jabusch HC. Musician's cramp as manifestation of maladaptive brain plasticity: arguments from instrumental differences. Ann N Y Acad Sci. 2012 Apr;1252:259-65. doi: 10.1111/j.1749-6632.2012.06456.x. PMID 22524368
- [Background] Schmidt A, Jabusch HC, Altenmuller E, Hagenah J, Bruggemann N, Hedrich K, Saunders-Pullman R, Bressman SB, Kramer PL, Klein C. Dominantly transmitted focal dystonia in families of patients with musician's cramp. Neurology. 2006 Aug 22;67(4):691-3. doi: 10.1212/01.wnl.0000230148.00035.f9. PMID 16924027
- [Background] Altenmuller E, Jabusch HC. Focal dystonia in musicians: phenomenology, pathophysiology, triggering factors, and treatment. Med Probl Perform Art. 2010 Mar;25(1):3-9. PMID 20795373
- [Background] Schuele S, Jabusch HC, Lederman RJ, Altenmuller E. Botulinum toxin injections in the treatment of musician's dystonia. Neurology. 2005 Jan 25;64(2):341-3. doi: 10.1212/01.WNL.0000149768.36634.92. PMID 15668436
- [Background] Pullman SL, Greene P, Fahn S, Pedersen SF. Approach to the treatment of limb disorders with botulinum toxin A. Experience with 187 patients. Arch Neurol. 1996 Jul;53(7):617-24. doi: 10.1001/archneur.1996.00550070055012. PMID 8929169
- [Background] Peterson DA, Berque P, Jabusch HC, Altenmuller E, Frucht SJ. Rating scales for musician's dystonia: the state of the art. Neurology. 2013 Aug 6;81(6):589-98. doi: 10.1212/WNL.0b013e31829e6f72. Epub 2013 Jul 24. PMID 23884039
- [Background] Chang FC, Frucht SJ. Motor and Sensory Dysfunction in Musician's Dystonia. Curr Neuropharmacol. 2013 Jan;11(1):41-7. doi: 10.2174/157015913804999531. PMID 23814536

RESULTS

PARTICIPANT FLOW:
Period: Cycle 1: Week 1-4
Arm/Group | Placebo Then Botulinum Toxin | Incobotulinumtoxin A Then Placebo
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Washout: Weakness Back to Baseline
Arm/Group | Placebo Then Botulinum Toxin | Incobotulinumtoxin A Then Placebo
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Cycle 2: Week 12-15
Arm/Group | Placebo Then Botulinum Toxin | Incobotulinumtoxin A Then Placebo
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Botulinum Toxin Then Placebo: Incobotulinumtoxin A dose first does then boosters at week 2 and week 4 then 4 weeks washout, then Placebo first dose, with boosters at 2 week and week 4.
- Total: Total of all reporting groups
Arm/Group | Placebo Then Botulinum Toxin | Botulinum Toxin Then Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Full Range); unit: years] | 52.68 [38.04 to 56.71] | 49.66 [37.76 to 63.00] | 50.2 [37.76 to 63.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Perception of Change - Blinded Rater 1
Description: The principal outcome measure was improvement in musical performance, measured by blinded rater, using physician global perception of change at post treatment compared to at 8 weeks. Categories are very much improved, much improved, minimal improved, no change, and minimal worse.
Time Frame: at visit 4 (week 8)
Population: Data not collected for one participant. Data results for Week 8 before crossover treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: matching placebo injection
- Incobotulinum Toxin Injection: Incobotulinumtoxin A used on average doses between 10U and 30 Units per subject, but at no time did any subject receive over 100 Units. Each study visit, the assessing physician selected the muscles and the amounts of medication to be injected.
Arm/Group | Placebo | Incobotulinum Toxin Injection
Number analyzed (Participants) | 11 | 9
Participants
  Very much improved | 1 | 1
  Much Improved | 1 | 4
  Minimally Improved | 3 | 3
  No Change | 3 | 0
  Minimally Worse | 3 | 1

2. Primary Outcome: Physician Global Perception of Change - Blinded Rater 2
Description: as for outcome 1
Time Frame: at visit 4 (week 8)
Population: Data not collected for one participant. Data results for Week 8 before crossover treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Incobotulinum Toxin Injection
Number analyzed (Participants) | 11 | 9
Participants
  Very much improved | 0 | 0
  Much Improved | 1 | 2
  Minimal Improved | 4 | 5
  No Change | 3 | 1
  Minimal Worse | 3 | 1

3. Primary Outcome: Rating of Overall Musical Performance - Blinded Rater 1
Description: Rating of overall musical performance based on comparison to baseline video at week 8.
  Rating from +3, very much improved to -3, very much worse. Higher score indicates more improvement.
Time Frame: baseline and at 8 weeks
Population: Data not collected for one participant. Data results for Week 8 before crossover treatment.
Measure: Count of Participants; unit: Participants
Groups:
- XEOMIN: Incobotulinumtoxin A used on average doses between 10U and 30 Units per subject, but at no time did any subject receive over 100 Units. Each study visit, the assessing physician selected the muscles and the amounts of medication to be injected.
Arm/Group | Placebo | XEOMIN
Number analyzed (Participants) | 11 | 9
Participants
  +3 Very much improved | 0 | 1
  +2 Much improved | 2 | 2
  +1 Minimally improved | 0 | 3
  0 No change | 5 | 2
  -1 Minimal worse | 4 | 1
  -2 Much worse | 0 | 0
  -3 Very much worse | 0 | 0

4. Primary Outcome: Rating of Overall Musical Performance - Blinded Rater 2
Description: Rating of overall musical performance based on comparison to baseline video at week 8.
  Best Overall Musical Performance on 7 point scale from +3 Very much improved to -3 Very much worse. Higher score indicates more improvement.
Time Frame: baseline and week 8
Population: Data not collected for one participant. Data results for Week 8 before crossover treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Incobotulinum Toxin Injection
Number analyzed (Participants) | 11 | 9
Participants
  +3 Very much improved | 0 | 0
  +2 Much Improved | 3 | 2
  +1 Minimally Improved | 0 | 4
  0 No Change | 5 | 2
  -1 Minimally Worse | 3 | 1
  -2 Much worse | 0 | 0
  -3 Very much worse | 0 | 0

5. Primary Outcome: Quantitative MIDI Analysis Comparison
Description: The principal outcome measure will be improvement in musical performance, measured by self-rated questionnaire, quantitative Musical Instrument Digital Interface (MIDI) analysis and blinded high speed video analysis post treatment compared to baseline and 24 weeks.
Time Frame: baseline at 24 weeks
Population: data not collected at 24 weeks
Arm/Group | Placebo | Incobotulinum Toxin Injection
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Blinded High Speed Video Analysis Comparison
Description: The principal outcome measure will be improvement in musical performance, measured by self-rated questionnaire, quantitative MIDI analysis and blinded high speed video analysis post treatment compared to baseline and 24 weeks.
Time Frame: baseline and at 24 weeks
Population: data not collected at 24 weeks
Groups:
- Incobotulinumtoxin A: Incobotulinumtoxin A used on average doses between 10U and 30 Units per subject, but at no time did any subject receive over 100 Units. Each study visit, the assessing physician selected the muscles and the amounts of medication to be injected.
Arm/Group | Placebo | Incobotulinumtoxin A
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Perceived Stress Scale (PSS)
Description: Patient reported outcomes measured by questionnaires that address adverse events and the impact of quality of life using the perceived stress scale. A 10-item questionnaire, each item scored 0 (never) to 4 (very often), full scale from 0-40, with higher score indicating higher perceived stress. the more often the person perceives stress Change in PSS at week 8 compared to baseline
Time Frame: baseline and at 8 weeks
Population: Data results for Week 8 before crossover treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | XEOMIN
Number analyzed (Participants) | 11 | 10
score on a scale | -1.429 (0.864) | -0.5031 (0.946)

8. Secondary Outcome: Change in Medical Research Council (MRC) Scale
Description: Motor strength using a dynamometer of the finger/wrist/elbow flexors to document any treatment induced weakness.
  Scale from 0-4, higher score indicates poorer health outcomes.
Time Frame: baseline and at 8 weeks
Population: Data results for Week 8 before crossover treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | XEOMIN
Number analyzed (Participants) | 11 | 10
score on a scale
  Right FDP dig 2 | 0.07 (0.0655) | -0.087 (0.0654)
  R Lumb dig 4 | -0.013 (0.0493) | -0.1190 (0.0492)

9. Secondary Outcome: Change in Motor Strength Comparison
Description: Motor strength tested using a dynamometer to document any weakness the treatment may produce as compared to the baseline visit and 8 weeks.
  Dynamometer (DYN) - is a mechanical device that measures the pounds of force that a muscle exerts, Grip - a device that measures grip strength, and finger flexors digit 2 and 3 (FF d2-3). These measures are the amount of lbs of force exert. The higher number is the highest exerted out of 3 tries.
Time Frame: baseline and at 8 weeks
Population: Data results for Week 8 before crossover treatment.
Measure: Least Squares Mean (Standard Error); unit: lbs of force exert
Arm/Group | Placebo | XEOMIN
Number analyzed (Participants) | 11 | 10
lbs of force exert
  DYN pnch 4 max | 0.679 (0.5954) | -3.037 (0.629)
  DYN pnch 4 avg | 1.065 (0.5688) | -2.323 (0.5951)
  DYN pnch 3 max | 0.5570 (0.7079) | -2.905 (0.7522)
  DYN pnch 3 Avg | 1.1440 (0.6354) | -2.2 (0.6762)
  Grip max | 3.084 (4.6889) | -25.04 (4.9933)
  Grip avg | 4.944 (4.721) | -22.172 (4.9974)
  FF D2-3 | 19.526 (7.1284) | -4.423 (6.5695)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Placebo | Incobotulinum Toxin Injection
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 12/20 | 7/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Incobotulinum Toxin Injection (N=21)
Weakness (Musculoskeletal and connective tissue disorders) | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT02107261/Prot_SAP_000.pdf